CLINICAL TRIAL: NCT01105390
Title: A Phase II Trial of AMG 102 in Combination With Pemetrexed and Cisplatin in Patients With Malignant Pleural Mesothelioma
Brief Title: AMG 102, Pemetrexed Disodium, and Cisplatin in Treating Patients With Malignant Pleural Mesothelioma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: withdrawn
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E1B09; NCI-2011-02068 (Registry Identifier: CTRP (Clinical Trials Reporting System)); U10CA021115 (NIH); CDR0000670445 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-01

CONDITIONS: Advanced Malignant Mesothelioma; Epithelial Mesothelioma; Recurrent Malignant Mesothelioma; Sarcomatous Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — rilotumumab; Cisplatin; Pemetrexed

ARMS (1):
- Treatment (rilotumumab, cisplatin, pemetrexed disodium) (Experimental): Patients receive anti-HGF monoclonal antibody AMG 102 (AMG 102) IV over 1 hour, pemetrexed disodium IV over 10 minutes, and cisplatin IV over 1 hour on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients without disease progression may continue AMG 102 IV over 1 hour on day 1, every 3 weeks, as maintenance therapy in the absence of disease progression.
  Interventions: Biological: rilotumumab; Drug: cisplatin; Drug: pemetrexed disodium; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: rilotumumab — Given IV
  Other Names: AMG 102; anti-HGF monoclonal antibody AMG 102
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: pemetrexed disodium — Given IV
  Other Names: ALIMTA; LY231514; MTA
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving AMG 102 together with pemetrexed disodium and cisplatin works in treating patients with malignant pleural mesothelioma. Monoclonal antibodies, such as AMG 102, can block tumor growth in different ways. Some block the ability of tumor cells to grow or spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as pemetrexed disodium and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving AMG 102 together with pemetrexed disodium and cisplatin may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the progression-free survival of patients with malignant pleural mesothelioma (MPM) treated with anti-HGF monoclonal antibody AMG 102 in combination with pemetrexed disodium and cisplatin.

SECONDARY OBJECTIVES:

I. To assess the toxicity associated with this regimen in these patients. II. To determine the response rate of patients treated with this regimen. III. To determine the overall survival of patients treated with this regimen. IV. To evaluate multiple potential correlative biomarkers in MPM that are relevant to this combined regimen, including serum HGF and mesothelin levels, c-met expression by IHC in tumor specimens, presence of c-met mutations in tumor, and the presence of thymidylate synthetase (TS) and excision repair cross complementing protein-1 (ERCC1) polymorphisms.

OUTLINE: This is a multicenter study.

Patients receive anti-HGF monoclonal antibody AMG 102 (AMG 102) IV over 1 hour, pemetrexed disodium IV over 10 minutes, and cisplatin IV over 1 hour on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients without disease progression may continue AMG 102 IV over 1 hour on day 1, every 3 weeks, as maintenance therapy in the absence of disease progression. Some patients undergo blood sample collection at baseline and periodically during study for correlative biomarker studies. Tumor samples from diagnostic tissue may also be analyzed.

After completion of study therapy, patients are followed up periodically every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and cytologically confirmed malignant mesothelioma of the pleura

  * All subtypes allowed
  * Disease not amenable to curative surgery
* Measurable disease

  * Patients with disease not measurable by standard RECIST criteria (i.e., pleural rinds/thickening only) allowed
  * Pleural effusions or positive bone scans are not considered measurable
* No prior radiotherapy to the target lesion or measurable lesion unless the site has subsequent evidence of progression
* Patients who have undergone pleurodesis allowed

  * Post-pleurodesis CT scan required
* No known or suspected brain metastases
* ECOG performance status 0-1
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 1.5 times ULN
* ALT and AST ≤ 1.5 times ULN
* Albumin ≥ 2.5 g/dL
* Creatinine clearance ≥ 45 mL/min OR serum creatinine ≤ 1.5 times ULN
* Able to take folic acid and vitamin B12
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must agree to use effective contraception
* No active infection or serious concomitant systemic disorder in compatible with the study
* No thrombosis or vascular ischemic events within the last 12 months, including any of the following:

  * Deep venous thrombosis
  * Pulmonary embolism
  * Transient ischemic attack
  * Cerebral infarction
  * Myocardial infarction
* No peripheral edema ≥ grade 3
* No serious or non-healing wounds
* No second primary malignancy except in situ carcinoma of the cervix or breast, other in situ malignancies, adequately treated basal cell carcinoma of the skin, or other malignancy within the past 3 years with no evidence of recurrence
* No concurrent antiretroviral therapy for HIV-positive patients
* At least 4 weeks since prior radiotherapy
* More than 30 days since major surgery procedures or > 14 days since any minor surgical procedure and recovered

  * Central venous catheter placement, fine-needle aspiration, thoracentesis, or paracentesis are not considered major or minor surgical procedures
* No prior systemic chemotherapy for mesothelioma
* No prior intracavity cytotoxic drugs or immunomodulators (unless for the purpose of pleurodesis)
* No prior anti-HGF monoclonal antibody AMG 102, other c-MET, or HGF inhibitors
* No prior or concurrent anticoagulation therapy within the past 7 days

  * Low-dose Coumadin-type anticoagulants or low-molecular weight heparin for prophylaxis against central venous catheter thrombosis allowed
* No investigational agents within the past 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From registration to clinical evidence of disease progression or death without progression, assessed up to 3 years

SECONDARY OUTCOMES:
Toxicity defined as a grade 4 hemorrhagic event or a grade 5 event | Up to 30 days after completion of study treatment
  Graded using the NCI CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: James Stevenson, Principal Investigator — Eastern Cooperative Oncology Group